CLINICAL TRIAL: NCT05060679
Title: Presepsin:Gelsolin Ratio, as a Promising Marker of Sepsis-related Organ Dysfunction: a Pilot Study
Brief Title: Presepsin:Gelsolin Ratio in Sepsis-related Organ Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dániel Ragán, MD, Principal Investigator, University of Pecs
Other Study IDs: 4327.316-2900/KK15/2011
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Acute Kidney Injury Due to Sepsis; Septic Shock; Acute Respiratory Distress Syndrome
Keywords: Sepsis-3; Organ dysfunction; Prognosis; Presepsin; Gelsolin; Presepsin:gelsolin ratio; Novel biomarker
MeSH Terms: conditions — Sepsis; Shock, Septic; Respiratory Distress Syndrome; Meretoja syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (Serum; Plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-sepsis: Non-septic patients receive supportive treatment at the ICU.
  Interventions: Other: Supportive therapy at the ICU
- Sepsis: Patients receive sepsis therapy.
  Interventions: Other: Sepsis therapy
- Sepsis-related organ dysfunction: Patients receive sepsis therapy and advanced supportive treatment based on the occurrence of specific sepsis-related organ dysfunctions.
  Interventions: Other: Sepsis-related organ dysfunction therapy

INTERVENTIONS:
Other: Supportive therapy at the ICU — Non-septic ICU patients received adequate supportive treatment (fluid resuscitation, respiratory, anticoagulation, antimicrobial and vasopressor therapy along with sedation, ulcer prophylaxis and nutrition. Blood sampling for non-septic patients were the first (T1) and third (T3) postoperative morning at the ICU. Besides, 23 healthy outpatients were documented without sepsis or sepsis-related organ dysfuntion as a control group.
  Groups: Non-sepsis
Other: Sepsis therapy — Patients receiving sepsis therapy followed the international guidelines of the 2016 Surviving Sepsis Campaign (SSC) regarding respiratory, antimicrobial, anticoagulation, vasopressor and hydrocortisone therapy, along with adequate fluid resuscitation, sedation, ulcer prophylaxis and nutrition. Blood samples were collected at the ICU from this patient group at three time points (T1-3): T1: within 12 hours after admission; T2: second day morning; T3: third day morning of follow-up.
  Groups: Sepsis
Other: Sepsis-related organ dysfunction therapy — Patient management of sepsis and sepsis-related organ dysfunction followed the international guidelines of the 2016 Surviving Sepsis Campaign (SSC) regarding respiratory, antimicrobial, anticoagulation, vasopressor and hydrocortisone therapy, along with adequate fluid resuscitation, sedation, ulcer prophylaxis, nutrition and renal replacement therapy (if needed). In this patient group, blood sampling was performed at three time points (T1-3): T1: within 12 hours after admission; T2: second day morning; T3: third day morning of follow-up.
  Groups: Sepsis-related organ dysfunction

SUMMARY:
In the present study, 126 patients were enrolled (23 control, 38 non-septic and 65 septic patients). Blood samples were collected from septic patients at the intensive care unit (ICU) at three time points (T1-3): T1: within 12h after admission; T2: second day morning; T3: third day morning. Sampling points for non-septic ICU patients were T1 and T3. Exclusion criteria were patients under 18 years of age, unobtainable consent, end-stage renal disease requiring chronic dialysis or kidney transplantation and patients with malignancies needing palliative care. Not more than one sample (venous blood) was collected from control patients. Plasma presepsin levels were determined by an automated chemiluminescence-based Point of Care instrument while serum gelsolin levels were measured using an automated immune turbidimetric assay. Plasma presepsin concentrations were expressed as pg/mL, while serum gelsolin levels were expressed as mg/L. Data were compared with laboratory and clinical parameters. Patients were categorized by the Sepsis-3 definitions and 10-day mortality data were investigated. Presepsin:gelsolin ratio was evaluated in major sepsis-related organ dysfunctions including hemodynamic disturbances, respiratory insufficiency and acute kidney injury (AKI).

DETAILED DESCRIPTION:
Presepsin is the 13-kDa soluble N-terminal fragment of the 55-kDa cluster of differentiation (CD) marker protein CD14, which is the receptor for lipopolysaccharide (LPS) and LPS-binding protein complexes. CD14 is a glycoprotein expressed mostly on the membrane surface of macrophages, monocytes and granulocytes which is released and degraded during inflammation after the recognition of pathogen-associated molecular patterns (PAMP), thus probably resulting in earlier elevation of plasma presepsin (PSEP) levels than the conventional sepsis biomarkers (C-reactive protein, procalcitonin). There is a growing body of evidence indicating increasing PSEP levels as kidney function decreases (e.g. during chronic kidney disease or sepsis-related AKI). Gelsolin (GSN) is a multifunctional protein existing in three different isoforms. Secreted or plasma GSN (MW = 83 kDa) is an essential component of the so-called extracellular actin scavenger system, therefore, decreasing serum GSN levels were reported in various clinical conditions (e.g. severe sepsis, multiple organ dysfunction syndrome (MODS), extensive trauma, acute liver failure, myocardial infarction). As albumin levels also tend to decrease in severe catabolic conditions, the simultaneous measurement of PSEP and GSN could prove to be useful regarding the diagnosis and prognosis of sepsis and sepsis-related organ dysfunction. Therefore, a new potential marker was investigated: the presepsin:gelsolin (PSEP:GSN) ratio. The main focuses of this study were analyzing the time course of PSEP:GSN ratio in non-septic and septic patients, while also investigating its diagnostic and prognostic utility in various sepsis-related organ dysfunctions in contrast to the conventional sepsis markers and clinical prognostic scores.

ELIGIBILITY:
Inclusion Criteria:

* Non-septic patients needing ICU supportive treatment after major surgical interventions
* Sepsis
* Sepsis-related organ dysfunction (e.g. acute kidney injury, hemodynamic instability, acute respiratory distress syndrome)

Exclusion Criteria:

* under 18 years of age
* unobtainable consent
* end-stage renal disease
* kidney transplantation
* malignancies needing palliative care

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy control individuals (n=23), non-septic ICU patients (n=38) and septic patients (n=65) were enrolled, while the septic group was also investigated based on the occurrence of sepsis-related organ dysfunction (e.g. acute kidney injury, hemodynamic instability, acute respiratory distress syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Plasma Presepsin concentrations | 3 days
  Plasma samples were centrifuged (10 min, 1500 g), then sample aliquots were stored without preservatives at -70 °C until analysis. Plasma presepsin levels were measured using an automated Point of Care instrument (PATHFAST; LSI Medience Corporation, Tokyo, Japan) based on a chemiluminescent enzyme immunoassay.
Serum gelsolin concentrations | 3 days
  Clotted blood samples were centrifuged (10 min, 1500 g), then sample aliquots were stored without preservatives at -70 °C until analysis. Serum gelsolin levels were determined with an automated immune turbidimetric assay (Cobas 8000/c502 module (Roche Diagnostics GmbH, Mannheim, Germany)).

SECONDARY OUTCOMES:
Presepsin:gelsolin ratios | 5 days
  Plasma presepsin levels were determined by an automated Point of Care instrument, while serum gelsolin concentrations were measured using an immune turbidimetric assay, therefore Presepsin:gelsolin ratios could be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Dániel Ragán, MD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Péter Kustán, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Zoltán Horváth-Szalai, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Balázs Szirmay, MD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Attila Miseta, MD, Dsc, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Gábor Woth, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs; Tamás Kőszegi, MD, PhD, Principal Investigator — Department of Laboratory Medicine, Medical School, University of Pécs; Diána Mühl, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Medical School, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ragan D, Kustan P, Horvath-Szalai Z, Szirmay B, Miseta A, Woth G, Koszegi T, Muhl D. Presepsin: gelsolin ratio, as a promising marker of sepsis-related organ dysfunction: a prospective observational study. Front Med (Lausanne). 2023 May 5;10:1126982. doi: 10.3389/fmed.2023.1126982. eCollection 2023. PMID 37215727